CLINICAL TRIAL: NCT02006446
Title: Are Sperm Head Vacuoles Associated With Sperm Nuclear Alterations?
Brief Title: Relationship Between Sperm Head Vacuoles and Sperm DNA Alterations in Infertile Men
Acronym: VATES
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/005/HP
Record Dates: First submitted 2013-11-25; First posted 2013-12-10 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Male Infertility
Keywords: Male infertility; sperm head vacuoles; sperm morphology; aneuploidy; DNA fragmentation; abnormal chromatin condensation; telomere abnormalities
MeSH Terms: conditions — Infertility, Male; Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — spermatozoa
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VATES: men with altered spermograms (isolated teratozoospermia or oligo-astheno-teratozoospermia)

SUMMARY:
In men presenting sperm alterations, the selection of genetically undamaged spermatozoa need to be improved in order to increase the success of assisted reproduction treatments.

The aim of this study is to determine whether the presence of sperm head vacuoles is associated with sperm DNA alterations.

DETAILED DESCRIPTION:
The use of intracytoplasmic sperm injection (ICSI) has greatly improved the treatment of severe male infertility, especially for men with oligo-astheno-teratozoospermia (OAT). This in vitro fertilization procedure allows the direct injection of a single spermatozoon into an oocyte. The sperm used for ICSI is selected under a microscope at a 400x magnification. Several studies have reported that de novo chromosomal abnormalities are increased in children born from ICSI , thereby raising the question of the genetic quality of spermatozoa used for ICSI.

A method called MSOME (high magnification Motile Sperm Organelle Morphology Examination), which allows the detailed morphological evaluation of motile spermatozoa in real time and under high magnification (6600x), was developed in 2001. With this technique, fine morphological abnormalities - mainly vacuoles in the head of spermatozoa - were detected. The use of MSOME for the detection of morphologically normal sperm for ICSI gave rise to a technique called IMSI (Intracytoplasmic Morphologically Selected sperm Injection). Higher pregnancy rates were obtained with IMSI compared to ICSI and sperm head vacuoles were found to negatively affect assisted reproduction success rates and embryo development. The use of IMSI also decreases the risk of sex chromosome aneuploidy in embryos .

Several authors found that the presence of large vacuoles in the sperm head correlates with several nuclear alterations: DNA fragmentation , abnormal chromatin condensation and aneuploidy . However, these studies are controversial and were performed on few spermatozoa. In order to improve the selection of spermatozoa with a normal chromosomal content, it is essential not only to confirm the existence of a relationship between sperm head vacuoles and altered sperm nuclear quality but also to better characterize these alterations.

The main goal of this study is to investigate the correlation between sperm head vacuole areas and sperm aneuploidy rates in men with isolated teratozoospermia or OAT. Vacuole areas will be measured by MSOME and aneuploidy rates by FISH for chromosomes 18, X and Y. Moreover, the correlation between sperm head vacuole areas and other nuclear alterations (DNA fragmentation, abnormal chromatin condensation, telomere abnormalities) will be evaluated. Semen samples from 200 patients recruited over a 2-year period will be collected, stored and analyzed.

This study involves the collection of relevant medical information. The computer website for the patient database is secure and protected by a password. The information will be entered and only be viewed by the investigators. On-site monitoring visits will be conducted throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* men
* 18 years old or more
* affiliated to social security
* with isolated teratozoospermia or oligo-astheno-teratozoospermia according to the WHO guidelines (2010):

  * sperm concentration < 15 million per ml or sperm number < 39 million per ejaculate
  * progressive motility < 35%
  * morphologically normal forms < 50% according to the modified David's classification (Auger et al., 2001
  * mobile spermatozoa selected by density gradient centrifugation > 1 million, in previous spermograms
* with normal constitutional karyotypes (46, XY)
* signed an informed consent

Exclusion Criteria:

* with abnormal constitutional karyotypes
* with a major alteration of sperm parameters, with mobile spermatozoa selected by density gradient centrifugation < 1 million
* under tutorship or guardianship by court order

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: infertile men attending the assisted reproduction units in Rouen and Lille
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between mean vacuole areas in sperm heads (measured by MSOME) and sperm aneuploidy rates for chromosomes X, Y and 18 (evaluated by FISH) | up to 30 months

SECONDARY OUTCOMES:
Total sperm count | 1 day
Percentage of mobile spermatozoa | 1 day
Percentage of morphologically abnormal spermatozoa | 1 day
Mean vacuole area threshold (measured with Receiver Operating Characteristic curves) | up to 30 months
Correlation coefficient between vacuole areas and sperm DNA fragmentation (evaluated by TUNEL analysis) | up to 30 months
Correlation coefficient between vacuole areas and abnormal chromatin condensation (evaluated by aniline blue staining) | up to 30 months
Correlation coefficient between vacuole areas and telomere number, distribution and length (evaluated by quantitative FISH) | up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Rives, MD., PhD., Principal Investigator — Laboratoire de Biologie de la Reproduction - CECOS - EA 4308, CHU - Hôpitaux de Rouen
Locations (2):
- France (2):
  - Laboratoire de spermiologie, CHRU de Lille, Hôpital Calmette CHRU de Lille
  - Laboratoire de Biologie de la Reproduction - CECOS - EA 4308, CHU - Hôpitaux de Rouen, Rouen

REFERENCES:
- [Background] Antinori M, Licata E, Dani G, Cerusico F, Versaci C, d'Angelo D, Antinori S. Intracytoplasmic morphologically selected sperm injection: a prospective randomized trial. Reprod Biomed Online. 2008 Jun;16(6):835-41. doi: 10.1016/s1472-6483(10)60150-2. PMID 18549694
- [Background] Auger J, Eustache F, Andersen AG, Irvine DS, Jorgensen N, Skakkebaek NE, Suominen J, Toppari J, Vierula M, Jouannet P. Sperm morphological defects related to environment, lifestyle and medical history of 1001 male partners of pregnant women from four European cities. Hum Reprod. 2001 Dec;16(12):2710-7. doi: 10.1093/humrep/16.12.2710. PMID 11726600
- [Background] Bartoov B, Berkovitz A, Eltes F. Selection of spermatozoa with normal nuclei to improve the pregnancy rate with intracytoplasmic sperm injection. N Engl J Med. 2001 Oct 4;345(14):1067-8. doi: 10.1056/NEJM200110043451416. No abstract available. PMID 11586970
- [Background] Bartoov B, Berkovitz A, Eltes F, Kogosovsky A, Yagoda A, Lederman H, Artzi S, Gross M, Barak Y. Pregnancy rates are higher with intracytoplasmic morphologically selected sperm injection than with conventional intracytoplasmic injection. Fertil Steril. 2003 Dec;80(6):1413-9. doi: 10.1016/j.fertnstert.2003.05.016. PMID 14667877
- [Background] Boitrelle F, Ferfouri F, Petit JM, Segretain D, Tourain C, Bergere M, Bailly M, Vialard F, Albert M, Selva J. Large human sperm vacuoles observed in motile spermatozoa under high magnification: nuclear thumbprints linked to failure of chromatin condensation. Hum Reprod. 2011 Jul;26(7):1650-8. doi: 10.1093/humrep/der129. Epub 2011 May 2. PMID 21536591
- [Background] Bonduelle M, Van Assche E, Joris H, Keymolen K, Devroey P, Van Steirteghem A, Liebaers I. Prenatal testing in ICSI pregnancies: incidence of chromosomal anomalies in 1586 karyotypes and relation to sperm parameters. Hum Reprod. 2002 Oct;17(10):2600-14. doi: 10.1093/humrep/17.10.2600. PMID 12351536
- [Background] Figueira Rde C, Braga DP, Setti AS, Iaconelli A Jr, Borges E Jr. Morphological nuclear integrity of sperm cells is associated with preimplantation genetic aneuploidy screening cycle outcomes. Fertil Steril. 2011 Mar 1;95(3):990-3. doi: 10.1016/j.fertnstert.2010.11.018. Epub 2010 Dec 4. PMID 21130987
- [Background] Foresta C, Garolla A, Bartoloni L, Bettella A, Ferlin A. Genetic abnormalities among severely oligospermic men who are candidates for intracytoplasmic sperm injection. J Clin Endocrinol Metab. 2005 Jan;90(1):152-6. doi: 10.1210/jc.2004-1469. Epub 2004 Oct 27. PMID 15509635
- [Background] Franco JG Jr, Baruffi RL, Mauri AL, Petersen CG, Oliveira JB, Vagnini L. Significance of large nuclear vacuoles in human spermatozoa: implications for ICSI. Reprod Biomed Online. 2008 Jul;17(1):42-5. doi: 10.1016/s1472-6483(10)60291-x. PMID 18616888
- [Background] Franco JG Jr, Mauri AL, Petersen CG, Massaro FC, Silva LF, Felipe V, Cavagna M, Pontes A, Baruffi RL, Oliveira JB, Vagnini LD. Large nuclear vacuoles are indicative of abnormal chromatin packaging in human spermatozoa. Int J Androl. 2012 Feb;35(1):46-51. doi: 10.1111/j.1365-2605.2011.01154.x. Epub 2011 Apr 28. PMID 21535011
- [Background] Garolla A, Fortini D, Menegazzo M, De Toni L, Nicoletti V, Moretti A, Selice R, Engl B, Foresta C. High-power microscopy for selecting spermatozoa for ICSI by physiological status. Reprod Biomed Online. 2008 Nov;17(5):610-6. doi: 10.1016/s1472-6483(10)60307-0. PMID 18983744
- [Background] Hazout A, Dumont-Hassan M, Junca AM, Cohen Bacrie P, Tesarik J. High-magnification ICSI overcomes paternal effect resistant to conventional ICSI. Reprod Biomed Online. 2006 Jan;12(1):19-25. doi: 10.1016/s1472-6483(10)60975-3. PMID 16454928
- [Background] Oliveira JB, Massaro FC, Baruffi RL, Mauri AL, Petersen CG, Silva LF, Vagnini LD, Franco JG Jr. Correlation between semen analysis by motile sperm organelle morphology examination and sperm DNA damage. Fertil Steril. 2010 Oct;94(5):1937-40. doi: 10.1016/j.fertnstert.2010.01.042. Epub 2010 Mar 2. PMID 20189558
- [Background] Perdrix A, Travers A, Chelli MH, Escalier D, Do Rego JL, Milazzo JP, Mousset-Simeon N, Mace B, Rives N. Assessment of acrosome and nuclear abnormalities in human spermatozoa with large vacuoles. Hum Reprod. 2011 Jan;26(1):47-58. doi: 10.1093/humrep/deq297. Epub 2010 Nov 18. PMID 21088015
- [Background] Van Steirteghem A, Bonduelle M, Devroey P, Liebaers I. Follow-up of children born after ICSI. Hum Reprod Update. 2002 Mar-Apr;8(2):111-6. doi: 10.1093/humupd/8.2.111. PMID 12099626
- [Background] Vanderzwalmen P, Hiemer A, Rubner P, Bach M, Neyer A, Stecher A, Uher P, Zintz M, Lejeune B, Vanderzwalmen S, Cassuto G, Zech NH. Blastocyst development after sperm selection at high magnification is associated with size and number of nuclear vacuoles. Reprod Biomed Online. 2008 Nov;17(5):617-27. doi: 10.1016/s1472-6483(10)60308-2. PMID 18983745
- [Background] Watanabe S, Tanaka A, Fujii S, Mizunuma H, Fukui A, Fukuhara R, Nakamura R, Yamada K, Tanaka I, Awata S, Nagayoshi M. An investigation of the potential effect of vacuoles in human sperm on DNA damage using a chromosome assay and the TUNEL assay. Hum Reprod. 2011 May;26(5):978-86. doi: 10.1093/humrep/der047. Epub 2011 Feb 28. PMID 21362682
- [Background] Wilding M, Coppola G, di Matteo L, Palagiano A, Fusco E, Dale B. Intracytoplasmic injection of morphologically selected spermatozoa (IMSI) improves outcome after assisted reproduction by deselecting physiologically poor quality spermatozoa. J Assist Reprod Genet. 2011 Mar;28(3):253-62. doi: 10.1007/s10815-010-9505-5. Epub 2010 Nov 12. PMID 21072684